CLINICAL TRIAL: NCT00451880
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL281 Administered Orally to Subjects With Solid Tumors
Brief Title: Study of XL281 in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Kanya Rajangam, MD/Senior Manager, Clinical Research, Exelixis, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL281-001
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Cancer; Non-small-cell Lung Cancer; Colorectal Cancer; Papillary Thyroid Cancer; Melanoma
Keywords: Cancer; Solid Tumors; NSCLC
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Thyroid Cancer, Papillary; Melanoma | interventions — Famotidine

ARMS (3):
- Arm 1 (Experimental): XL281 administered once a day
  Interventions: Drug: XL281
- Arm 2 (Experimental): XL281 administered twice a day
  Interventions: Drug: XL281
- Arm 3 (Experimental): XL281 administered once a day. Subjects in this arm will be dosed under fed conditions, fasted conditions, and with a concomitant single dose of 40 mg famotidine, during the second, third, and fourth week of the first cycle.
  Interventions: Drug: XL281; Drug: famotidine

INTERVENTIONS:
Drug: XL281 — Gelatin capsules supplied as 5-, 25-, and 100-mg strengths
Drug: famotidine — single dose, supplied as 20-mg or 40-mg tablets
  Other Names: Pepcid®
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine the safest dose of the multiple Raf kinase inhibitor (including c-Raf, B-Raf, and the activated mutant B-RafV600E) XL281, how often it should be taken, and how well subjects with cancer tolerate XL281. This study will also determine how the body reacts to XL281 when it is taken with and without food, and with and without Pepcid (famotidine), a drug that inhibits stomach acid production.

ELIGIBILITY:
Key Inclusion Criteria:

* The subject has a histologically confirmed solid tumor that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective, and there are no therapies known to prolong survival. Subjects treated at the MTD (once- or twice- daily) must have a diagnosis of colorectal cancer, non-small-cell lung cancer (no longer recruiting), melanoma, or papillary thyroid cancer. Certain other eligibility requirements must also be met.
* The subject is ≥18 years old.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* The subject has adequate organ and marrow function.
* The subject is capable of understanding the protocol and has signed the informed consent document.
* Sexually active subjects (male and female) must use medically acceptable methods of contraception during the course of the study and for 3 months after study drug discontinuation.
* Female subjects of childbearing potential must have a negative pregnancy test at screening.
* The subject has had no other diagnosis of malignancy (unless non-melanoma skin cancer, carcinoma in situ of the cervix, or a malignancy diagnosed ≥5 years ago, and has had no evidence of disease for 5 years prior to screening for this study).
* The subject must meet certain other eligibility requirements.

Key Exclusion Criteria:

* The subject has received anticancer treatment (eg, chemotherapy, radiotherapy, cytokines, or hormones) within 28 days (6 weeks for nitrosoureas or mitomycin C) before the first dose of study drug.
* The subject has received treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within a certain amount of time before the first dose of study drug.
* The subject has received any other investigational agent within 28 days of first dose of XL281.
* The subject has not recovered to Grade ≤1 from adverse events (AEs) or to within 10% of baseline values due to investigational or other agents administered more than 30 days prior to study enrollment. Some irreversible toxicities from previous treatment may be allowed.
* The subject requires treatment with antacids (continual treatment), proton pump inhibitors, or H2 receptor antagonists.
* The subject has a primary brain tumor or known brain metastases.
* The subject has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* The subject is pregnant or breastfeeding.
* The subject is known to be positive for the human immunodeficiency virus (HIV).
* The subject has an allergy or hypersensitivity to components of the XL281 formulation or to famotidine.
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
* The subject is receiving anticoagulation with warfarin or coumarin-related compounds (low-dose warfarin ≤ 1 mg/day, heparin, and low-molecular weight heparin are permitted)
* The subject must meet certain other eligibility requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose (MTD) of once daily or twice daily oral administration of XL281 | Assessed at periodic visits
To assess the pharmacokinetic/pharmacodynamic/preliminary clinical activity relationship following XL281 administration in different tumor types from subjects treated at the MTD | Assessed at periodic visits
To determine the bioavailability of XL281 under fed and fasted conditions, and with or without the concomitant use of a single dose of famotidine in subjects with solid tumors | Assessed during the second, third, and fourth week of the first cycle of dosing

SECONDARY OUTCOMES:
Plasma pharmacokinetics of once daily or twice daily oral administration of XL281 | Assessed at periodic visits

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas